CLINICAL TRIAL: NCT03866785
Title: Physical Activity Experiment on Male Prostate Cancer Patients : Feasibility Multicenter Study of an Innovative Follow-up by Peers
Brief Title: Physical Activity Experiment on Male Prostate Cancer Patients
Acronym: ACTI_PAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18CH034; 2018-A00710-55 (Other: ANSM)
Record Dates: First submitted 2018-10-22; First posted 2019-03-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cancer Prostate
Keywords: Prostate cancer; Physical activity; Activity actigraph; Peer; Program; Sports medicine
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study is composed of 3 dependent steps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STEP 1: Patient with prostate cancer (Other): First, patients with prostate cancer will be included during step 1. They will have an interview.
  Interventions: Diagnostic Test: interview
- STEP 2: Patient with prostate cancer and a physical activity (Other): Secondly, patient with prostate cancer and a physical activity will be included during step 2. They are called "peer".
  They will have a questionnaire Adult Physical Activity Questionnaire (APAQ), an activity actigraph and a peer training. The peer will help patients to realize the Physical Activity Program during step 3.
  Interventions: Diagnostic Test: Adult Physical Activity Questionnaire (APAQ); Device: Activity actigraph; Other: Peer training
- STEP 3: Physical Activity Program (Other): Finally, patients with prostate cancer (different from step 1) and who agrees to participate at the Physical Activity Program will be included during step 3.
  They will have an activity actigraph and a questionnaire Adult Physical Activity Questionnaire (APAQ) at inclusion and 3 months later.
  They will receive the Physical Activity Program.
  Interventions: Diagnostic Test: Adult Physical Activity Questionnaire (APAQ); Device: Activity actigraph; Other: Physical Activity Program

INTERVENTIONS:
Diagnostic Test: interview — The goal is to evaluate the needs, the constraints and representations of patients on the practice of physical activity.
  Arms: STEP 1: Patient with prostate cancer
Diagnostic Test: Adult Physical Activity Questionnaire (APAQ) — The goal of this questionnaire is to evaluate the sedentary lifestyle of patients.
  Arms: STEP 2: Patient with prostate cancer and a physical activity; STEP 3: Physical Activity Program
Device: Activity actigraph — An activity actigraph will use by the patient for a week. It measures the level of physical activity and the sedentary lifestyle of patients.
  Arms: STEP 2: Patient with prostate cancer and a physical activity; STEP 3: Physical Activity Program
Other: Peer training — The goal of the peer training will organize once a week for 3 weeks for a patient.
  After this training, they will have :
  * Skills in physical activity advice
  * Knowledge of functional signs (symptoms)
  * Knowledge to examine heart rate and perceived effort rate
  Arms: STEP 2: Patient with prostate cancer and a physical activity
Other: Physical Activity Program — During the Physical Activity Program, patients will be supervised by peers and a clubs and sports associations labeled sport-health by Olympic and Sports Committee of the Loire Department.
  The peer will coach the patient once a week minimum for 3 months.
  Arms: STEP 3: Physical Activity Program

SUMMARY:
Prostate cancer is the most common cancer in France (56,841 cases in 2012). Although the benefits of physical activity (PA) in cancer patients are currently well established in the scientific literature, several studies have shown that this population is not sufficiently active. Strengthen patient adherence to prevention counseling by the physical activity (PA) is emerging as a new challenge for personalized treatment in oncology. In order to encourage the engagement and maintenance in a regular PA of cancer patients, first, their experiences of physical activity (PA) practice should be considered and their initial social representations of the practice considered. Secondarily, it is also important to identify health professionals who retain a key role in defining the framework, objectives and means of action to promote lifestyle changes towards a more active lifestyle. In addition, peer mentoring appears to offer promising perspectives for promoting adherence and long-term maintenance in physical activity (PA) of cancer patients.

DETAILED DESCRIPTION:
The main objective of this project is to measure the adherence of prostate cancer patients to a physical activity program with a tracking of the motivation by a pair.

ELIGIBILITY:
Inclusion Criteria for patient in step1, 2 and 3:

* Major patient followed for prostate cancer:

  * located or locally advanced,
  * metastatic and / or resistant to castration and chemotherapy.
* Cancer diagnosed at least 1 year ago
* Patient affiliated or beneficiary to social security
* Signed informed consent.

In more, step 2 = Patient with Physical Activity for at least 1 year

Exclusion Criteria:

For step 1= In the course of cancer treatment (excluding hormonal therapy)

For step 2= Patient in sedentary lifestyle

For step 3=

* In the course of cancer treatment (excluding hormonal therapy)
* Cardiac or respiratory conditions contraindicating physical activity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Physical Activity sessions performed | At month 3
  Analysis of the proportion (%) of Physical Activity sessions performed after 3 months of intervention.

SECONDARY OUTCOMES:
physical activity via activity actigraph | At month 3
  Assessment of physical activity via activity actigraph
sedentary lifestyle via activity actigraph | At month 3
  Assessment of sedentary lifestyle via activity actigraph
Patient's activation | At month 3
  Measure patient's activation via questionnaire Patient Activation Measure (PAM).
brakes blocking intervention | At month 3
  Identification of brakes blocking intervention via interviews and Adult Physical Activity Questionnaire (APAQ). APAQ measures the sleeping time (h/night), sedentary time (h/week) and physical activity time (h/day)
levers favoring intervention | At month 3
  Identification of levers favoring intervention via interviews and Adult Physical Activity Questionnaire (APAQ). APAQ measures the sleeping time (h/night), sedentary time (h/week) and physical activity time (h/day)
Peers mobilized | At month 3
  Number of peers mobilized

CONTACTS AND LOCATIONS:
Overall Officials: David HUPIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU Saint-Etienne, Saint-Etienne
  - ICLN - département de radiothérapie, Saint-Priest-en-Jarez
  - ICLN - Oncologie médicale, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No